CLINICAL TRIAL: NCT06491810
Title: Oxygen Saturation in the Leg Musculature Affected by Peripheral Arterial Disease During Exercise on an Arm Ergometer
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Nove de Julho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marilia de Almeida Correia, PhD, University of Nove de Julho
Other Study IDs: EBPAD_StO
Record Dates: First submitted 2024-06-27; First posted 2024-07-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Arterial Disease
Keywords: Exercise; Oxygen saturation; Intermittent Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity; Intermittent Claudication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arm crank exercise: The exercise session will consist of 15 sets of 2 minutes of exercise in arm ergometer with an intensity equivalent to 13-15 on the Borg's perceived exertion scale.
  Interventions: Other: Arm crank exercise

INTERVENTIONS:
Other: Arm crank exercise — The arm ergometer exercise will be the only intervention implemented during the study.

SUMMARY:
Studies with arm ergometer (AE) training have shown benefits in the functional capacity of patients with peripheral arterial disease (PAD) bypassing the main barrier to exercise in these patients, pain during walking exercise. The only study that proposed to investigate the mechanism involved in this adaptation observed that chronically training with EB promoted improvement in the oxygen saturation (StO₂) of the leg muscles during walking. However, how arm exercise could improve leg muscle StO₂ remains unknown.

The goal of this study is to analyze what happens during AE on the tissue oxygen saturation (StO₂) of the leg affected by PAD.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 50 years;
2. with PAD confirmed by clinical diagnosis and ankle-brachial index (ABI) < 0.90 in one or both limbs;
3. experiencing symptoms of intermittent claudication (IC) during walking;
4. with a body mass index (BMI) not exceeding 30 kg/m²;
5. with medical clearance to participate in the project;
6. presenting calf skinfold thickness less than 20 mm due to interference of adiposity with the light penetration of the NIRS probe and finger oxygen saturation > 95% to ensure that impaired pulmonary gas exchange does not affect the calf oxygen saturation measurements.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral artery disease
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Calf Muscule Oxygen Saturation (%) | Just before, during 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 minutes of exercise, and after 10 minutes of exercise.
  The parameters of calf muscle oxygenation will be collected using the non-invasive Near-Infrared Spectroscopy (NIRS) technique, with an NIRS spectrometer and a dedicated laptop computer. The NIRS sensor will be placed on the calf region, on the leg with the lower ankle brachial index, at the level of the largest calf circumference. The equipment will be programmed for continuous recording throughout the experimental session, covering the pre-exercise, during exercise with arm ergometer, and post-exercise periods.

SECONDARY OUTCOMES:
Oxyhemoglobin (micromol) | Just before, during 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 minutes of exercise, and after 10 minutes of exercise.
  The parameters of calf muscle oxygenation will be collected using the non-invasive Near-Infrared Spectroscopy (NIRS) technique, with an NIRS spectrometer and a dedicated laptop computer. The NIRS sensor will be placed on the calf region, on the leg with the lower ankle brachial index, at the level of the largest calf circumference. The equipment will be programmed for continuous recording throughout the experimental session, covering the pre-exercise, during exercise with arm ergometer, and post-exercise periods.
Deoxyhemoglobin (micromol) | Just before, during 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 minutes of exercise, and after 10 minutes of exercise.
  The parameters of calf muscle oxygenation will be collected using the non-invasive Near-Infrared Spectroscopy (NIRS) technique, with an NIRS spectrometer and a dedicated laptop computer. The NIRS sensor will be placed on the calf region, on the leg with the lower ankle brachial index, at the level of the largest calf circumference. The equipment will be programmed for continuous recording throughout the experimental session, covering the pre-exercise, during exercise with arm ergometer, and post-exercise periods.
Total hemoglobin (micromol) | Just before, during 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 minutes of exercise, and after 10 minutes of exercise.
  The parameters of calf muscle oxygenation will be collected using the non-invasive Near-Infrared Spectroscopy (NIRS) technique, with an NIRS spectrometer and a dedicated laptop computer. The NIRS sensor will be placed on the calf region, on the leg with the lower ankle brachial index, at the level of the largest calf circumference. The equipment will be programmed for continuous recording throughout the experimental session, covering the pre-exercise, during exercise with arm ergometer, and post-exercise periods.
Subjective perception of exertion (score) | During 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 minutes of exercise.
  Subjective perception of effort will be assessed using the Borg Scale, from 6 to 20, where participants rate their perceived exertion during the exercise session.
Pain (score) | During 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 minutes of exercise.
  Pain will be assessed using the Visual Analog Scale (VAS), where participants mark their current level of pain on a horizontal line typically 10 centimeters in length. One end represents "no pain," while the other end signifies "worst pain imaginable."

CONTACTS AND LOCATIONS:
Overall Officials: Jéssika Silva, Ms, Study Chair — University of Nove de Julho
Locations (1):
- University Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cavalcante BR, Ritti-Dias RM, Soares AH, Lima AH, Correia MA, De Matos LD, Gobbi F, Leicht AS, Wolosker N, Cucato GG. A Single Bout of Arm-crank Exercise Promotes Positive Emotions and Post-Exercise Hypotension in Patients with Symptomatic Peripheral Artery Disease. Eur J Vasc Endovasc Surg. 2017 Feb;53(2):223-228. doi: 10.1016/j.ejvs.2016.11.021. Epub 2016 Dec 21. PMID 28012910